CLINICAL TRIAL: NCT04360603
Title: The Safety Outcomes of 27 Gauge Vitrectomy for Posterior Segment Disease in High Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201907025RINB
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Wound Complication; High Myopia; Vitrectomy
Keywords: vitrectomy; high myopia; wound leakage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 27 gauge system (Experimental): study group, using 27G vitrectomy system
  Interventions: Device: 27G
- 25 gauge system (Active Comparator): control group, using 25G vitrectomy system
  Interventions: Device: 25G

INTERVENTIONS:
Device: 27G — using 27G vitrectomy system to perform standard transconjunctival sutureless vitrectomy
  Arms: 27 gauge system
Device: 25G — using 25G vitrectomy system to perform standard transconjunctival sutureless vitrectomy
  Arms: 25 gauge system

SUMMARY:
In recent decade, a major improvement in vitreoretinal surgery was the use of small gauge surgical systems that improved the safety of vitrectomy and also reduced the surgical time. However, there were still some concerns regarding small gauge vitrectomy system, especially 27-gauge system, in the stability of its instruments and the efficacy of removing vitreous during surgery. Although there were some studies that had reported the surgical outcomes of 27G vitrectomy system, none had focused on patients with high myopia. The highly myopic patients usually had thinner sclera, which was a risk factor for wound leakage after sutureless vitrectomy, they also had longer axial length which would make the surgical procedure more difficult especially in macular surgery.

Based on previous clinical finding, gas leakage was 36.4% in 25G , while 27G sclerotomy showing less leakage comparing to larger gauge sclerotomy, the investigators believe 27G may have its clinical advantages in overcoming the thinner sclera of high myopia, and show the superiority of leakage control.

Hypothesis:

The 27G vitrectomy system has lower sclerotomy wound leakage rate compared with 25G system

ELIGIBILITY:
Inclusion criteria:

1. Highly myopic patients (axial length 26~31mm)
2. Diagnosed with vitreoretinal pathology that require vitrectomy
3. Never received vitrectomy before

Exclusion criteria:

1. Surgical planning including scleral buckling during operation
2. Surgical planning including combined phacoemulsification
3. Surgical planning including the use of silicone oil and/or perfluorocarbon liquid
4. Previous ocular surgery involving conjunctival manipulation and scarring such as pterygium removal/trabeculectomy
5. Previous vitrectomy
6. Previous ocular trauma involving corneal/corneoscleral/scleral/conjunctival full thickness laceration
7. Medical history with known connective tissue disease(s)
8. Age younger than 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative sclerotomy site wound leakage | immediately at the end of surgery
  The incidence of intraoperative sclerotomy site wound leakage

SECONDARY OUTCOMES:
Incidence of postoperative sclerotomy site wound leakage | post-operation day 1, 3, week 1, month 1, 3, 6
  postoperative complication
Incidence of hypotony | post-operation day 1, 3, week 1, month 1, 3, 6
  intraoperative and postoperative complication
Incidence of endophthalmitis | post-operation day 1, 3, week 1, month 1, 3, 6
  postoperative complication
Incidence of instrument bending | during operation
  intraoperative complications
Incidence of subconjunctival hemorrhage | post-operation day 1, 3, week 1, month 1, 3, 6
  postoperative complication

OTHER OUTCOMES:
total vitrectomy time | during operation
  total vitrectomy time
total surgical time | during operation
  total surgical time
visual outcomes | post-operation month 1, 3, 6
  best-corrected visual acuity and visual acuity changes
Incidence of anatomical success | post-operation month 1, 3, 6
  anatomical success, such as restoration of normal foveal contour, reattachment of retina

CONTACTS AND LOCATIONS:
Overall Officials: Chung-May Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No